CLINICAL TRIAL: NCT05574985
Title: A Randomized, Open, Positive Controlled Clinical Study to Evaluate the Immunogenicity and Safety of Recombinant Omicron-Delta COVID-19 Vaccine (CHO Cell) in People Aged 18 Years and Over
Brief Title: Recombinant Omicron-Delta COVID-19 Vaccine (CHO Cell)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LKM-2022-DO-NCV-01
Record Dates: First submitted 2022-10-10; First posted 2022-10-12 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: COVID-19
Keywords: Recombinant Vaccine; Omicron-Delta
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Research Group (Experimental): People 6 to 15 months after the completion of basic immunization with inactivated COVID-19 vaccine were vaccinated one dose of the study vaccine
  Interventions: Biological: Recombinant Omicron-Delta COVID-19 Vaccine (CHO Cell)
- Control Group (Active Comparator): People 6 to 15 months after the completion of basic immunization with inactivated COVID-19 vaccine were vaccinated with one dose of control vaccine
  Interventions: Biological: Inactivated COVID-19 vaccine (Vero Cell)
- Observation group ① (Experimental): People 6 to 9 months after the completion of the inactivated COVID-19 vaccine booster immunization were vaccinated one dose of the study vaccine
  Interventions: Biological: Recombinant Omicron-Delta COVID-19 Vaccine (CHO Cell)
- Observation group ② (Experimental): People 6 to 15 months after the completion of basic immunization with COVID-19 recombinant vaccine were vaccinated one dose of the study vaccine
  Interventions: Biological: Recombinant Omicron-Delta COVID-19 Vaccine (CHO Cell)

INTERVENTIONS:
Biological: Recombinant Omicron-Delta COVID-19 Vaccine (CHO Cell) — Injected one dose of research vaccine
  Arms: Observation group ①; Observation group ②; Research Group
Biological: Inactivated COVID-19 vaccine (Vero Cell) — Injected one dose of control vaccine
  Arms: Control Group

SUMMARY:
Popular topic:A Clinical Study of Recombinant Omicron-Delta COVID-19 Vaccine (CHO Cell) Overall design:The study was designed as a randomized, open and controlled study.

Study population: People aged 18 years and above and 6-15 months after the completion of basic immunization or 6-9 months after the completion of enhanced immunization with the new coronal prototype vaccine.

Test groups:Study group；Control group；Observation group ①；Observation group ②

DETAILED DESCRIPTION:
Research topic: A randomized, open, positive controlled clinical study to evaluate the immunogenicity and safety of the recombinant novel coronavirus protein vaccine (CHO cell) of Omicron-Delta strain in people aged 18 years and above.

Product name:Recombinant Omicron-Delta COVID-19 Vaccine (CHO Cell),each dose contains 25μg DO-RBD protein/0.5mL/bottle.

Indications: Prevention of respiratory diseases caused by new coronavirus infection.

Research purpose:

Main purpose:To evaluate the immunogenicity of Omicron Delta strain recombinant novel coronavirus protein vaccine (CHO cells) against new crown variants (Delta, Omicron BA. 2，Omicron BA. 5) in people aged 18 years and above.

Secondary objectives: To evaluate the safety of recombinant novel coronavirus protein vaccine (CHO cells) of Omicron Delta strain in people aged 18 years and above.

Research design:The study adopted a randomized, open and controlled design. Study group and control group: 150 patients who completed the basic immunization with inactivated new crown vaccine were randomly divided into study group and control group, and were injected with study vaccine and control vaccine respectively; Observation group ①: 75 patients who completed homologous booster immunization with inactivated new coronal vaccine were injected with one dose of study vaccine; Observation group ②: 75 patients who completed the basic immunization of new coronal recombinant vaccine were injected with one dose of study vaccine.

Safety endpoint:

1. Incidence of all AEs occurring within 28 days after vaccination:(1)Total incidence of AEs;(2) Incidence of AEs associated with the investigational vaccine;(3) Incidence of AEs of Grade 3 or above;(4) Incidence of AEs associated with the investigational vaccine of Grade 3 or above;(5) Incidence of AEs resulting in withdrawal;(6)Incidence of AEs resulting in withdrawal that are associated with the investigational vaccine;
2. Incidence of all serious adverse events (SAEs) within six months after vaccination, and incidence of vaccine-related SAEs.

Immunogenicity endpoint:

1. Primary end point:

   GMT of neutralizing antibody in the serum of subjects against the SARS-CoV-2 Delta, BA.2, and BA.5 within 14 days after vaccination.
2. Secondary end points:GMT of neutralizing antibody in the serum of subjects of the study group and the control group against SARS-CoV-2 Delta, BA.2, BA. 5 within six months after vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the Informed Consent, he was 18 years old or above;
2. Normal body temperature (axillary temperature < 37.3 ℃/oral temperature < 37.5 ℃);
3. Meet one of the following conditions: 1) 6-15 months after the basic immunization (2 injections) of the inactivated vaccine of the prototype strain of COVID-19-19 has been completed; 2) 6-9 months after the booster immunization (3 injections) of the inactivated vaccine of the prototype strain of COVID-19 has been completed; 3) 6-15 months after basic immunization (3 injections) of recombinant vaccine of COVID-19 prototype strain has been completed.
4. The vaccines used to complete the above basic immunization or enhanced immunization were produced by Beijing Biotech, Wuhan Biotech, Sinovac and Zhifeilong Koma, and the same kind of vaccine was inoculated throughout the whole process.
5. Female subjects over 18 years old were not pregnant (blood pregnancy test was negative), were not in lactation and took effective contraceptive measures within 4 weeks after inoculation; The male subject must agree to take effective contraceptive measures by himself and his partner within 4 weeks after signing the informed consent and vaccination.
6. Subjects have the ability to understand the research procedure, voluntarily sign the informed consent form after informed consent, can comply with the requirements of the clinical research protocol, and can and is willing to complete the entire required research plan.

Exclusion Criteria:

1. A history of serious allergy to any vaccine in the past, or a history of serious allergy to any component of the studied vaccine, including aluminum preparations, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, dyspnea, angioneurotic edema, allergic constitution (such as allergic to two or more drugs, food or pollen);
2. Confirmed cases of novel coronavirus infection, asymptomatic infections or positive history of novel coronavirus nucleic acid testing;
3. Patients with uncontrollable lymphoproliferative disease, aplastic anemia, primary immune thrombocytopenia (ITP), and haemorrhagic disease;
4. A history of congenital or acquired immunodeficiency or autoimmune diseases;
5. The life expectancy of patients with malignant tumors is less than 1 year;
6. Patients with uncontrolled epilepsy and other progressive nervous system diseases (such as transverse myelitis, Guillain Barre syndrome, demyelinating disease, etc.);
7. Patients with acute disease, or acute attack period of chronic disease, or uncontrolled severe chronic disease, such as hypertension beyond the control of drugs (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
8. Those who have received inactivated vaccine within one week or attenuated vaccine within four weeks before vaccination;
9. Subjects who have participated in other clinical studies or are participating in other clinical studies within 3 months;
10. The investigator believes that the subject has any disease or condition that may put the subject at risk, that the subject cannot complete the study as required by the protocol, and that there are conditions that interfere with the evaluation of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-10-09 (Actual); Study Completion 2023-03-18 (Actual)

PRIMARY OUTCOMES:
Immunogenicity end point 1 | 14 days after vaccination
  Blood samples were collected from subjects on the 14th day after vaccination, and serum was obtained after centrifugation. Then, the geometric mean titer (GMT) of neutralizing antibodies against COVID-19 variants (Delta, Omicron BA.2，Omicron BA.5) was obtained from the serum samples of subjects on the 14th day after vaccination.
Safety end point 1 | 28 days after vaccination
  The contact card was recovered on the 28th day after vaccination, and the clinician determined whether there was an adverse event and entered it into the EDC system. After statistical analysis, the incidence of all adverse events within 28 days was determined.
Safety end point 2 | 6 months after vaccination
  At the end of 6 months after vaccination, through telephone follow-up, the clinician learned whether the subject had serious adverse events, entered the information into the EDC system, and determined the incidence of all serious adverse events within 6 months through statistical analysis.

SECONDARY OUTCOMES:
Immunogenicity end point 4 | 6 months after vaccination
  Blood samples were collected from subjects at the end of 6 months after vaccination, and serum was obtained after centrifugation. Then, the geometric mean titer (GMT) of neutralizing antibodies against COVID-19 variants (Delta, Omicron BA.2，Omicron BA.5) was obtained from the serum samples of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, Professor, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No